CLINICAL TRIAL: NCT05504122
Title: Comparison of Laparoscopic Totally Extraperitoneal (TEP) and Lichtenstein Technique in Long-term Follow-up
Brief Title: Comparison of Laparoscopic Totally Extraperitoneal (TEP) and Lichtenstein Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Yuksel, Head of Gastroenterological Surgery, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOU KAEK 2012/161-17/14
Record Dates: First submitted 2022-07-31; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Hernia, Inguinal
Keywords: hernia; laparoscopic; Lichtenstein
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Totally Extraperitoneal (TEP) (Active Comparator): Patients who underwent Laparoscopic Totally Extraperitoneal (TEP) will be included in this group.
  Interventions: Procedure: inguinal hernia repair
- Open tension-free mesh repair technique (Lichtenstein) (Placebo Comparator): Patients with open tension-free inguinal hernia(Lichtenstein) repair will be included in this group.
  Interventions: Procedure: inguinal hernia repair

INTERVENTIONS:
Procedure: inguinal hernia repair — Patients who will undergo inguinal hernia repair will be divided into two groups(TEP versus Lichtenstein) according to the technique to be applied

SUMMARY:
Open tension-free mesh repair (Lichtenstein) and laparoscopic totally extraperitoneal (TEP) repair are the most commonly preferred techniques for inguinal hernia surgery. There's still a debate going on about which of these two techniques (open versus laparoscopic) is effective. This prospective randomized study aimed at comparing the early and long-term results of these two techniques (TEP vs. Lichtenstein).

DETAILED DESCRIPTION:
Various studies comparing the laparoscopic totally extraperitoneal (TEP) and Lichtenstein techniques have been reported. These studies have shown that TEP repair is associated with less postoperative pain and faster recovery. However, there are different views on the long-term (recurrence, chronic pain, etc.) results of the two techniques. This study was designed to compare the short- and long-term outcomes of open tension-free mesh repair technique(Lichtenstein) and laparoscopic repair technique(TEP).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with inguinal hernia (primary, recurrent, unilateral, bilateral)
* American Society of Anesthesiologists (ASA) score of I and II
* Gave informed consent to participate in the study

Exclusion Criteria:

* Patients with scrotal, strangulated, or obstructed hernia
* Periumbilical or subumbilical incision scar (median, right or left paramedian)
* Undergoing prostatectomy or abdominal bladder surgery
* Pfannenstiel incision scar
* ASA score >3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative complication status | up to the first 10 days postoperatively
  number of patients with complications
early period complication status | up to the first 3 months postoperatively
  number of patients with complications
late period complication status | Postoperative 3rd to 84th month
  number of patients with complications
early recurrence rate | up to the first 3 months postoperatively
  number of patients with recurrence
late recurrence rate | Postoperative 3rd to 84th month
  number of patients with recurrence

SECONDARY OUTCOMES:
Visual Analog Score for pain | postoperative 24th hour
  Units on a Scale; 0: no pain, 1-3: mild pain, 4-6: moderate pain, 7-9: severe pain, 10: worst pain possible.
total analgesic requirement | postoperative 1 to 10 days
  the number of analgesics used.
time to return to work after surgery | Postoperative 3rd month
  day
early complication status | postoperative 1st month
  Number of patients with complications

CONTACTS AND LOCATIONS:
Overall Officials: Murat Coskun, MD, Study Director — Kocaeli Derince Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langeveld HR, van't Riet M, Weidema WF, Stassen LP, Steyerberg EW, Lange J, Bonjer HJ, Jeekel J. Total extraperitoneal inguinal hernia repair compared with Lichtenstein (the LEVEL-Trial): a randomized controlled trial. Ann Surg. 2010 May;251(5):819-24. doi: 10.1097/SLA.0b013e3181d96c32. PMID 20395851
- [Background] Eklund AS, Montgomery AK, Rasmussen IC, Sandbue RP, Bergkvist LA, Rudberg CR. Low recurrence rate after laparoscopic (TEP) and open (Lichtenstein) inguinal hernia repair: a randomized, multicenter trial with 5-year follow-up. Ann Surg. 2009 Jan;249(1):33-8. doi: 10.1097/SLA.0b013e31819255d0. PMID 19106673
- [Background] O'Reilly EA, Burke JP, O'Connell PR. A meta-analysis of surgical morbidity and recurrence after laparoscopic and open repair of primary unilateral inguinal hernia. Ann Surg. 2012 May;255(5):846-53. doi: 10.1097/SLA.0b013e31824e96cf. PMID 22470068